CLINICAL TRIAL: NCT03678441
Title: A Feasibility Study of Electronic Neurocognitive Screening Tools in Surgery
Brief Title: Electronic Neurocognitive Tools in Screening for Mental Capability in Patients Undergoing Liver Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2018-0093; NCI-2018-01895 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0093 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-09-18; First posted 2018-09-19 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Liver and Intrahepatic Bile Duct Disorder
MeSH Terms: conditions — Digestive System Diseases | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (BrainCheck and paper and pen cognitive assessment) (Experimental): Patients receive the BrainCheck cognitive assessment over 15 minutes followed by the paper and pen assessment 2 months prior to surgery and within 2 months after surgery.
  Interventions: Behavioral: BrainCheck Cognitive Assessment; Procedure: Cognitive Assessment
- Group II (pen and paper and BrainCheck cognitive assessment) (Active Comparator): Patients receive the paper and pen assessment followed by the BrainCheck cognitive assessment over 15 minutes 2 months prior to surgery and within 2 months after surgery.
  Interventions: Behavioral: BrainCheck Cognitive Assessment; Procedure: Cognitive Assessment

INTERVENTIONS:
Behavioral: BrainCheck Cognitive Assessment — Receive BrainCheck cognitive assessment
  Other Names: BrainCheck
Procedure: Cognitive Assessment — Receive pen and paper cognitive assessment

SUMMARY:
This trial studies how well electronic neurocognitive tools work in screening for mental capability in patients who are undergoing liver surgery. Using electronic neurocognitive screening tools may help to better assess mental impairment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate feasibility of the electronic batteries, measured by the completion rate and time to completion of the batteries.

SECONDARY OBJECTIVES:

I. Comparison of the completion rate and time to completion between the written and electronic batteries.

II. Comparison of the scoring distribution between the screening tools.

EXPLORATORY OBJECTIVES:

I. Assess if a history of mental or cognitive illness or ongoing treatment with neuropsychiatric medications impact the ability to complete written and/or electronic neurocognitive screening.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive the BrainCheck cognitive assessment over 15 minutes followed by the paper and pen cognitive assessment within 2 months prior to surgery and within 2 months after surgery.

GROUP II: Patients receive the paper and pen cognitive assessment followed by the BrainCheck cognitive assessment over 15 minutes 2 months prior to surgery and within 2 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* All English-speaking patients undergoing hepatectomy at main campus University of Texas (UT)-MD Anderson Cancer Center who are cognitively able to provide informed consent in the opinion of the attending physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-08-17 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Completion rate of the BrainCheck battery | Up to 1 year
  Will be calculated along with a 95% confidence interval (CI).
Completion rate of the pen and paper assessment | Up to 1 year
  Will be calculated along with a 95% CI.
Average time to complete the BrainCheck battery | Up to 1 year
  Will be calculated along with a 95% CI.
Average time to complete the pen and paper assessment | Up to 1 year
  Will be calculated along with a 95% CI.
Difference in completion rate between the BrainCheck battery and paper and pen assessment | Up to 1 year
  Will be calculated along with 95% CIs.
Difference in time to completion between the BrainCheck battery and the pen and paper assessment | Up to 1 year
  Will be calculated along with 95% CIs.
Difference in score between the BrainCheck battery and the pen and paper assessments | Up to 1 year
  Will be calculated along with 95% CIs.
Sensitivity, specificity, negative predictive value, positive predictive value, and accuracy of the electronic battery compared to the validated St. Louis University Mental Status Examination (SLUMS) | Up to 1 year
  Will be calculated along with 95% CIs.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Newhook, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org